CLINICAL TRIAL: NCT04113239
Title: Study of the Genome, Gut Metagenome and Lifestyle of Patients With Incident Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Atlas Biomed (Industry)
Responsible Party: Sponsor
Other Study IDs: T2D+FFQ/GPAQ/Genome/Metagenome
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2; Metagenome; Genetic Predisposition
Keywords: Gut Metagenetics; Diabetes Mellitus, Type 2; Genetics; Microbiome; FFQ; GPAQ
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed Type 2 Diabetes Mellitus: Patients with incident type 2 diabetes mellitus
  Interventions: Diagnostic Test: 16S rRNA gene sequencing; Genetic: DNA-microarray genotyping
- Control: Volunteers without diagnosed type 2 diabetes mellitus and who don't meet the exclusion criteria
  Interventions: Diagnostic Test: 16S rRNA gene sequencing; Genetic: DNA-microarray genotyping

INTERVENTIONS:
Diagnostic Test: 16S rRNA gene sequencing — Taking a stool sample for gut microbiome DNA sequencing
Genetic: DNA-microarray genotyping — Taking a saliva sample for genotyping

SUMMARY:
A case-control study to identify microbiome and genetic differences between healthy people and patients with incident type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Two groups of people, one composed of healthy volunteers and the other of patients with incident type 2 diabetes mellitus who never received treatment for their condition, fill in the food frequency questionnaire and the physical activity questionnaire. DNA microarray genotyping is used to process the DNA samples of the participants. The data on the composition of the participants' gut microbiota is obtained through sequencing of their stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of incident type 2 diabetes mellitus

Exclusion Criteria:

* Hypoglycaemic therapy prescribed for the correction of any type of hyperglycaemia
* Diabetic ketoacidosis
* Inflammatory bowel diseases (ulcerative colitis, Crohn's disease, coeliac disease)
* Rheumatoid arthritis
* Tuberculosis
* Acute gastrointestinal conditions
* Irritable bowel syndrome
* Multiple intestinal polyposis
* Gallstone disease
* Acute pancreatitis
* Oncological diseases
* Serious mental disorders
* Recent (< 6 months) antimicrobial therapy
* Recent (< 3 months) proton pump inhibitors therapy
* Recent (< 3 months) surgical intervention
* Recent (< 3 weeks) use of probiotics, prebiotics, antacids, nonsteroidal anti-inflammatory drugs
* Pregnancy or breastfeeding
* Current alcohol/drug abuse or addiction within 12 months prior to screening
* Planned relocation from the study area during the study
* Other somatic pathologies or any factors that prevent the inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with incident type 2 diabetes mellitus from Russia, Moscow
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
HbA1C | Baseline
  Glycated hemoglobin level
Glucose | Baseline
  Fasting blood glucose level
Gut microbiome composition of participants | Baseline
  Bacteria abundance obtained via sequencing the DNA extracted from the stool sample
Genotypes of participants | Baseline
  Genotypes of thousands of SNPs obtained via DNA-microarray genotyping of the DNA extracted from the saliva sample

SECONDARY OUTCOMES:
Physical activity questionnaire | Baseline
  Physical Activity Questionnaire. It collects information on physical activity comprising 16 questions grouped in four domains: activity at work (1), travel to and from places (2), recreational activities (3), sedentary behaviour (4).
Food frequency questionnaire | 12 months before baseline
  Food frequency questionnaire assesses usual intake and portion size of more than 130 foods and beverages and more than 25 dietary supplements for the last 12 months. Responses are evaluated and analysed to compile a nutritional picture for each group of subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- City Clinical Hospital V.P. Demikhova, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No